CLINICAL TRIAL: NCT04054089
Title: Evaluating Inflammatory and Immunological Changes of HIV-positive Patients Switching to DTG Dual Regimen Compared to Those Switching to a Triple Drugs Regimen (B/F/TAF)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cristina Mussini (Other)
Responsible Party: Sponsor-Investigator, Cristina Mussini, Principal Investigator, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEBATE; 2018-003458-26 (EudraCT Number)
Record Dates: First submitted 2019-08-02; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir; Emtricitabine; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination; dolutegravir; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): B/F/TAF
  Interventions: Drug: Bictegravir 50 MG / Emtricitabine 200 MG / Tenofovir Alafenamide 25 MG [Biktarvy]
- B (Active Comparator): DTG+3TC
  Interventions: Drug: dolutegravir 50 mg / lamivudine 300 mg

INTERVENTIONS:
Drug: Bictegravir 50 MG / Emtricitabine 200 MG / Tenofovir Alafenamide 25 MG [Biktarvy] — Biktarvy OD
  Arms: A
Drug: dolutegravir 50 mg / lamivudine 300 mg — DTG +3TC (Dovato OD)
  Arms: B

SUMMARY:
Long-term side effects of antiretrovirals (ART) have led to the introduction in clinical practice of NRTI-sparing regimens as double- or mono- therapy and their use is now recommended in specific populations by International Guidelines. Indeed, based on the monitoring of surrogate markers of ART efficacy, most of these unconventional regimens, when used in switch studies, have shown to have a non-inferior virological efficacy and a good CD4 recovery compared to standard triple drug-based therapy.

At present, the best marker to evaluate the risk of developing of non-AIDS related events has not been determined. Interestingly, the analysis of the data of the investigator's and others cohorts have shown that, in contrast with recent data from ART-CC collaboration, a low CD4/CD8 ratio is a predictor of non-AIDS related events independently from CD4 cell count, while other studies have shown an association of this marker with non-AIDS defining cancers or, more recently, with pulmonary emphysema. Aim of the present study is to compare CD8 and CD4/CD8 slopes in patients switching with an undetectable viral load to the 2 regimens which will be more frequently used in clinical practice: i.e B/F/TAF and dolutegravir + lamivudine. Indeed, B/F/TAF is already a recommended regimen in all guidelines while dolutegravir + lamivudine is widely used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age = 18 years
2. The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
3. Patients infected by HIV-1
4. Patients under the first-line cART regimen with three antiretrovirals
5. HIV-RNA <=50 copies/mL for at least 12 months
6. No previous virological failures/blips
7. A female subject is eligible to enter the study if it is confirmed that she is:

   * Not pregnant or nursing
   * Of non-childbearing potential (e.g., women who have had a hysterectomy, have had both ovaries removed or medically documented ovarian failure, or are postmenopausal women >54 years of age with cessation for =12 months of previously occurring menses)
   * Of chilbearing potential and agrees to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following discontinuation of study drugs
   * Female subjects who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
8. Male subjects must agree to utilize a highly effective method of contraception (as defined in Appendix 5) during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 30 days following the last study drug dose.
9. Male subjects must agree to refrain from sperm donation from first dose until at least 30 days after the last study drug dose.

Exclusion Criteria:

1. Patients with chronic hepatitis B
2. Pregnant or breastfeeding women
3. Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
4. Known hypersensitivity to B/F/TAF FDC tablets, DTG and 3TC, their metabolites, or formulation excipient
5. Subjects receiving ongoing therapy with any of the following medications in the table below, including drugs not to be used with B, F, TAF, DTG and 3TC.

   Administration of any of the previous medications must be discontinued at least 30 days prior to the Day 1 visit and for the duration of the study
6. Documented resistance to any of the study drugs
7. Active, serious infection (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1.
8. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with protocol requirements. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
CD8 slope and consequent CD4/CD8 ratio difference between the 2 arms | week48

REFERENCES:
- [Derived] Cossarizza A, Cozzi-Lepri A, Mattioli M, Paolini A, Neroni A, De Biasi S, Tartaro DL, Borella R, Fidanza L, Gibellini L, Beghetto B, Roncaglia E, Nardini G, Milic J, Menozzi M, Cuomo G, Digaetano M, Orlando G, Borghi V, Guaraldi G, Mussini C. Evaluating immunological and inflammatory changes of treatment-experienced people living with HIV switching from first-line triple cART regimens to DTG/3TC vs. B/F/TAF: the DEBATE trial. Front Immunol. 2023 Oct 16;14:1279390. doi: 10.3389/fimmu.2023.1279390. eCollection 2023. PMID 37908359